CLINICAL TRIAL: NCT01260233
Title: The Effect of a Perioperative Smoking Cessation Program on Rates of Smoking Cessation/Reduction and Perioperative Complications: a Randomized Clinical Trial.
Brief Title: Effect of a Perioperative Smoking Cessation Program on Smoking Cessation/Reduction and Perioperative Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Philip Jones, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: R-10-476; 17342 (Other: UWO Health Sciences Research Ethics Board)
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Smoking; Tobacco Use
Keywords: smoking cessation; complications; cigarettes; preoperative; perioperative; surgery; education; nicotine replacement therapy
MeSH Terms: conditions — Smoking; Tobacco Use; Smoking Cessation | interventions — Nicotine; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No intervention. Patients will receive standard of care.
- Smoking cessation program (Experimental): Receives smoking cessation program
  Interventions: Other: Smoking cessation program

INTERVENTIONS:
Other: Smoking cessation program — Smoking cessation program includes:
  * brief smoking cessation counselling by preadmission nurse (less than 5 minutes)
  * smoking cessation brochures
  * referral to the Smokers' Helpline telephone advice line, run by the Canadian Cancer Society
  * free transdermal nicotine replacement therapy for 6 weeks Smokers of 10 cigarettes per day or more receive 4 weeks of nicoderm 21mg/day, 1 week of 14mg/day and 1 week of 7mg/day Smokers of less than 10 cigarettes per day receive 4 weeks of nicoderm 14mg/day and 2 weeks of 7mg/day
  Other Names: nicoderm; transdermal nicotine replacement therapy; nicotine replacement patch
  Arms: Smoking cessation program

SUMMARY:
The purpose of this study is to determine whether a perioperative smoking cessation program, implemented at least 3 weeks prior to elective surgery, is effective in increasing rates of smoking cessation or reduction. Intraoperative and immediate postoperative complications will also be compared.

DETAILED DESCRIPTION:
Previous studies have shown that patients have up to one-third fewer complications after surgery when they quit smoking at least several weeks before surgery. Nicotine replacement therapy (which relieves cravings for cigarettes) and support by healthcare professionals have been shown to help patients quit smoking, particularly when encountering a major health event (e.g. surgery). In addition, quitting smoking in preparation for surgery sometimes results in quitting for a longer period of time after surgery, giving these patients the health benefits of long-term smoking cessation such as reduced rates of cancer and heart disease.

The preadmission clinic at St. Joseph's Health Care, London, Ontario, is assessing how effective a new 'Stop Smoking' program is for patients preparing for surgery. The program will include brief counselling in the clinic, smoking cessation brochures, six weeks of free transdermal nicotine replacement therapy and a referral to the Canadian Cancer Society's Smokers' Helpline telephone advice line. Patients that are smokers and preparing for their elective surgery will be invited to join the study, then be assigned to a group that either participates in the program or not. These groups will then be compared in terms of success at quitting smoking and complication rates around the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* smokers (defined as those that smoke at least 2 cigarettes per day and have smoked within the last 7 days)
* over age 18
* presenting to preadmission clinic at St. Joseph's Health Care at least 3 weeks prior to scheduled date of surgery

Exclusion Criteria:

* less than age 18
* poor proficiency in English language
* pregnant
* breastfeeding
* unable to consent due to severe mental illness or dementia
* actively participating in another smoking cessation trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
smoking cessation | date of surgery
  Smoking cessation is defined as exhaled carbon monoxide (CO) of equal to or less than 7ppm on the day of surgery.

SECONDARY OUTCOMES:
smoking cessation/reduction | day of surgery
  Smoking cessation/reduction by self-report. Smoking cessation defined as zero cigarettes in the 7 days before surgery (but exhaled CO > 7ppm) Reduction defined as 50% or less of initial self-report.
Intraoperative complications and immediate post-operative complications | day of surgery
  Events occurring in the operating room or post-anesthetic care unit (PACU) as reported by a blinded anesthesiologist or blinded PACU nurse:
  Cardiovascular complications, Respiratory complications, Other (detailed description exceeds character limits)
Time until PACU readiness for discharge / actual time in PACU | day of surgery
  The time of arrival in PACU until the time the patient is deemed ready for discharge in accordance with hospital routine scoring system. The actual time spent in PACU (arrival until discharge) will also be compared.
  Patients bypassing PACU (e.g. patients having only sedation transferred directly from the operating room to surgical daycare prior to discharge home) will be considered separately.
Unanticipated hospital admission | day of surgery
  Patient booked as one-day stay, but later admitted to inpatient ward.
Hospital length of stay | until hospital discharge
  For inpatients only, the time from admission to surgical daycare until the patient is discharged home from the hospital.
Smoking cessation at 12 months | 1 year
  Self-reported smoking zero cigarettes in the 7 days prior to phone call. Phone call will occur at any time during the 12th month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Jones, MD, FRCPC, Principal Investigator — Western University, Canada
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Derived] Lee SM, Landry J, Jones PM, Buhrmann O, Morley-Forster P. Long-term quit rates after a perioperative smoking cessation randomized controlled trial. Anesth Analg. 2015 Mar;120(3):582-587. doi: 10.1213/ANE.0000000000000555. PMID 25695576